CLINICAL TRIAL: NCT03358238
Title: Modeling Mood Course to Detect Markers of Effective Adaptive Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Michigan (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: K01MH112876 (NIH); K01MH112876 (NIH); HUM00126732 (Other: University of Michigan); 2017-1322 (Other: University of Wisconsin)
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No weekly review (Placebo Comparator): Individuals will not review self-report and activity tracker data with an interviewer on a weekly basis over the phone.
  Interventions: Other: No weekly review
- Weekly review (Experimental): Individuals will review self-report and activity tracker data with an interviewer on a weekly basis over the phone.
  Interventions: Behavioral: Weekly review

INTERVENTIONS:
Behavioral: Weekly review — Each week in the study, an interviewer will review manic and depressive symptoms self-reported by a participant and patterns of activity, sleep, and heart rate collected by the participant's activity tracker.
  Arms: Weekly review
Other: No weekly review — An interviewer will not review self-report symptoms and patterns collected from an activity tracker.
  Other Names: Placebo
  Arms: No weekly review

SUMMARY:
The goal of this study is to learn how to engage individuals with bipolar disorder in long-term monitoring of daily patterns of mood, stress, sleep, circadian rhythm, and medical adherence. Knowledge gained will be used to develop a mobile health platform for the translation of a psychosocial intervention for bipolar disorder into an effective adaptive intervention.

DETAILED DESCRIPTION:
Bipolar disorder is a chronic illness of profound shifts in mood ranging from mania to depression. Bipolar disorder is successfully treated by combining medication with psychosocial therapy, but care can prove inadequate in practice. With gaps in coverage and medication, along with imprecise guidelines on when, where, and how to intervene, promising psychosocial therapies require adaptive strategies to better address the specific needs of individuals in a timely manner. To accomplish this, however, requires evidence-based practices for adapting a psychosocial therapy. The long-term goal of this study is to address this knowledge gap, by establishing a mobile health platform for translating a psychosocial therapy in bipolar disorder into an effective adaptive intervention.

An important first step and the specific goal of this study is to answer the question of how to engage individuals with bipolar disorder in long-term monitoring of their daily patterns of mood, stress, sleep, circadian rhythm, and medical adherence. To answer this question, individuals with bipolar disorder will interact with a smart-phone application and activity tracker over six weeks. Individuals will record their symptoms twice-daily with the smart-phone application while activity, sleep, and heart rate are recorded with their activity tracker. In addition, individuals will be interviewed on a weekly basis. The study focuses on testing three engagement strategies: using activity trackers rather than self-reports; reviewing recorded symptoms with another person on a weekly basis; and synthesizing a person's data into charts and graphs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with bipolar disorder
* Individuals with a smart-phone

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Cochran, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Til K, McInnis MG, Cochran A. A comparative study of engagement in mobile and wearable health monitoring for bipolar disorder. Bipolar Disord. 2020 Mar;22(2):182-190. doi: 10.1111/bdi.12849. Epub 2019 Oct 25. PMID 31610074
- [Derived] Cochran A, Belman-Wells L, McInnis M. Engagement Strategies for Self-Monitoring Symptoms of Bipolar Disorder With Mobile and Wearable Technology: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 May 10;7(5):e130. doi: 10.2196/resprot.9899. PMID 29748160

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were enrolled and subsequently excluded before the start of the study. One of these individuals died between the consent date and the start of the study, and the other was lost to follow-up between the consent date and study start.
Period: Overall Study
Arm/Group | No Weekly Review | Weekly Review
Started | 23 | 25
Completed | 23 | 24
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Weekly Review | Weekly Review | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (11.2) | 41.0 (10.6) | 41.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 19 | 22 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 19 | 22 | 41
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 47
Diagnosis [Number; unit: participants] — Number of participants per bipolar diagnostic category. Participants were diagnosed using the Diagnostic Interview for Genetic Studies (DIGS)26 with diagnoses reviewed by two clinicians after initial evaluation and reevaluated when suspected to change based on a clinically relevant event.
  participants
    Bipolar I | 17 | 16 | 33
    Bipolar II | 6 | 6 | 12
    Bipolar NOS | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Report They Are More Likely to Use a Smart-phone App Over an Activity Tracker to Monitor Their Symptoms
Description: Likelihood of using app over activity tracker is measured using a survey designed specifically for this study to evaluate participant engagement in monitoring symptoms. The relevant question asks 'Which are you more likely to use to monitor your symptoms' and has two mutually-exclusive options for an answer: 'An activity tracker' or 'A smart-phone app'. Engagement survey is conducted over the phone by an interviewer.
Time Frame: Study end (6 weeks)
Population: The analysis population includes both arms (rather than reporting outcomes by arm). Goals of this study went beyond measuring arm effects. Here, the question of interest is across the sample, do individuals prefer self-reporting over using an activity tracker. It is not of interest to know if the intervention changes this preference.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- All Participants: All participants from both arms of the study were asked the same question regarding their symptom-monitoring preference.
Arm/Group | All Participants
Number analyzed (Participants) | 47
proportion of participants | 0.404 [0.264 to 0.557]
Statistical Analysis 1: Comparison: All Participants; Test type: Other; Proportion = 0.404, 95% CI 2-sided [0.264 to 0.557] — Type of confidence interval = Clopper-Pearson

2. Primary Outcome: Average Proportion of Study Days With At Least 50% Completion of Daily Self-Reports Questions
Description: For each individual, adherence rate for self-reporting symptoms is measured/defined as the proportion of study days with at least 50% completion of of daily self-reports questions (i.e. 6 questions completed out of a total of 12).
  This measure is the average adherence rate for individuals in each of the two intervention arms: individuals who review their data with an interviewer ('Weekly review' arm) vs those who do not review their data with an interviewer ('No weekly review' arm).
Time Frame: Study end (6 weeks)
Measure: Mean (95% Confidence Interval); unit: proportion of study days
Groups:
- Review Arm: Individuals who reviewed weekly data with an interviewer
- No Review Arm: Individuals who did not review weekly data with an interviewer
Arm/Group | Review Arm | No Review Arm
Number analyzed (Participants) | 24 | 23
proportion of study days | 0.8185 [0.6954 to 0.9415] | 0.8168 [0.6865 to 0.9470]
Statistical Analysis 1: Comparison: Review Arm vs No Review Arm; Null hypothesis was that the difference in average adherence rates of self-reporting between arms was zero; Test type: Superiority; p = 0.99, t-test, 2 sided — Statistical significance was an alpha level of 0.05; Two-sample t test. Degrees of freedom = 45; Difference in Average Proportions = .0017, 95% CI 2-sided [-0.1774 to 0.1807] — Two-sample t confidence intervals

3. Primary Outcome: Average Proportion of Study Days With At Least 12 Hours of Activity Tracking
Description: For each individual, adherence rate for activity tracking is measured as the proportion of study days with at least 12 hours of activity tracking.
  This measure is the average adherence rates among individuals in either arm: individuals who review their data weekly with an interviewer ('Weekly review' arm) compared to individuals who do not review their data weekly with an interviewer ('No weekly review' arm)
Time Frame: Study end (6 weeks)
Measure: Mean (95% Confidence Interval); unit: proportion of study days
Arm/Group | Review Arm | No Review Arm
Number analyzed (Participants) | 24 | 23
proportion of study days | 0.7688 [0.6323 to 0.9054] | 0.7878 [0.6376 to 0.9379]
Statistical Analysis 1: Comparison: Review Arm vs No Review Arm; Null hypothesis was that the difference in average adherence rates to activity tracking between arms was zero; Test type: Superiority; p = 0.85, t-test, 2 sided — Statistical significance was considered an alpha level of 0.05; Two-sample t-test. Degrees of freedom = 45; Risk Difference (RD) = -0.0189, 95% CI 2-sided [-0.2215 to 0.1837] — Two-sample t confidence intervals

4. Primary Outcome: Proportion of Participants Who Have Higher Adherence Rates for Self-reporting Symptoms Than Adherence Rates for Activity Tracking
Description: For each individual, adherence rate for activity tracking is measured as the proportion of study days with at least 12 hours of activity tracking, whereas adherence rate for self-reporting symptoms is measured as the proportion of study days with at least 50% of daily self-reports survey questions completed.
Time Frame: Study end (6 weeks)
Population: For an individual, adherence rate for self-report is proportion of days with at least 50% completion of self-report questions; adherence rate for activity tracking is proportion of days with at least 12 hours of activity tracking.
  Participants with no difference in adherence rates between self-report and activity tracking were excluded.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Review Arm Participants With Unequal Adherence: Participants who reviewed weekly data with an interviewer and whose adherence rates were unequal for the self-report method of symptom monitoring compared to the activity tracker method.
- No Review Arm Participants With Unequal Adherence: Participants who did not review weekly data with interviewer and whose adherence rates for self-report and activity tracking differed
Arm/Group | Review Arm Participants With Unequal Adherence | No Review Arm Participants With Unequal Adherence
Number analyzed (Participants) | 21 | 18
Proportion of participants | 0.6667 [0.4303 to 0.8541] | 0.3889 [0.1730 to 0.6425]
Statistical Analysis 1: Comparison: Review Arm Participants With Unequal Adherence vs No Review Arm Participants With Unequal Adherence; Estimating proportion of individuals with higher adherence rates for self-report over activity tracking among individuals with unequal adherence rates; Test type: Other; Proportion = 0.5385, 95% CI 2-sided [0.3718 to 0.6991] — Type of confidence interval = Clopper-Pearson
Statistical Analysis 2: Comparison: Review Arm Participants With Unequal Adherence vs No Review Arm Participants With Unequal Adherence; Null hypothesis is that among individuals with unequal adherence rates, the proportion of individuals with greater adherence to self-report over activity tracking in the Review Arm is equal to the proportion of individuals with greater adherence to self-report over activity tracking in the No Review Arm; Test type: Superiority; p = 0.0828, Chi-squared; Degrees of freedom = 1

5. Secondary Outcome: Average Change From Baseline in Severity of Manic Symptoms, as Measured With the Young Mania Rating Scale
Description: The Young Mania Rating Scale consists of clinician-rated 11 items to evaluate symptoms of mania, such as elevated mood, energy, and irritability. Item scores are added together to get a total score, ranging from 0 to 60. A higher score indicates more severe manic symptoms.
Time Frame: Baseline, study end (6 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Review Arm | No Review Arm
Number analyzed (Participants) | 24 | 23
score on a scale | 0.67 [-0.54 to 1.88] | 0.91 [-1.32 to 3.15]
Statistical Analysis 1: Comparison: Review Arm vs No Review Arm; One participant had a single item missing on the Young Mania Rating Scale administered at study start. A zero was imputed for the missing item to recover a total score. Null hypothesis was that the average change in total scores was zero; Test type: Other; p = 0.20, t-test, 2 sided — Statistical significance was considered an alpha level of 0.05; One-sample t-test. Degrees of freedom = 46; Mean Difference (Net) = 0.79, 95% CI 2-sided [-0.42 to 1.99] — One participant had a single item missing on the Young Mania Rating Scale administered at study start. A zero was imputed for the missing item to recover a total score. One-sample t confidence intervals

6. Secondary Outcome: Average Change From Baseline in Severity of Depressive Symptoms, as Measured With the 17-item Structured Interview Guide for the Hamilton Rating Scale for Depression
Description: The 17-Item Structured Interview Guide for the Hamilton Rating Scale for Depression consists of 17 clinician-rated items to evaluate symptoms of depression, such as guilt, fatigue, and depressed mood. Item scores are summed to get a total score, ranging from 0 to 52. Higher scores indicate more severe symptoms.
Time Frame: Baseline, study end (6 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Review Arm | No Review Arm
Number analyzed (Participants) | 24 | 23
score on a scale | 0.67 [-2.07 to 3.40] | 1.13 [-1.43 to 3.69]
Statistical Analysis 1: Comparison: Review Arm vs No Review Arm; Null hypothesis was that average change in scores on the structured interview guide for the Hamilton rating scale for depression is zero; Test type: Other; p = 0.32, t-test, 2 sided — Statistical significance was considered an alpha level of 0.05; One-sample t test. Degrees of freedom = 46; Mean Difference (Net) = 0.89, 95% CI 2-sided [-0.91 to 2.70] — One-sample t confidence intervals

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of six weeks for each individual participant.
Arm/Group | No Weekly Review | Weekly Review
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/24
Other Adverse Events (participants affected / at risk) | 1/23 | 2/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Weekly Review (N=23) | Weekly Review (N=24)
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Participant was hospitalized for manic symptoms from 2/05/2018 to 2/12/2018, went to ER while experiencing manic symptoms on 2/24/2018, and was hospitalized again for manic symptoms from 2/26/2018 to 3/5/2018.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Weekly Review (N=23) | Weekly Review (N=24)
Fitbit Band Issue (Product Issues) | 1 (1) | 1 (1) — Issue with fit of activity tracker. Participants who indicated that their Fitbit did not fit properly returned the ill-fitting tracker and received a new one.
Participant Discontinuation (Product Issues) | 0 (0) | 1 (1) — Participant discontinued study due to discomfort with wearing Fitbit.
Missed Interviews (Social circumstances) | 1 (1) | 0 (0) — Participant missed Week 5, 6, & 7 interviews. Participant completed week 7 interview outside of +/- 1 day window to complete their study participation

LIMITATIONS AND CAVEATS:
Results regarding passive activity tracking may not generalize to other forms of passive tracking. Small sample sizes. Not powered to examine individual differences in responses to engagement survey at study end.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT03358238/Prot_SAP_000.pdf